CLINICAL TRIAL: NCT04613674
Title: A Multicentre, Randomized, Double-blind, Parallel-controlled Phase Ⅲ Study to Evaluate Camrelizumab Plus Chemotherapy vs Placebo Plus Chemotherapy as Neoadjuvant Therapy in Patients With Early or Locally Advanced Triple Negative Breast Cancer (TNBC).
Brief Title: A Study of Camrelizumab Plus Chemotherapy vs Placebo Plus Chemotherapy as Neoadjuvant Therapy in Participants With Triple Negative Breast Cancer (TNBC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR1210-III-322
Record Dates: First submitted 2020-10-29; First posted 2020-11-03 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — camrelizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Drug: Camrelizumab Plus Chemotherapy
- Arm B (Experimental)
  Interventions: Drug: placebo+chemotherapy

INTERVENTIONS:
Drug: Camrelizumab Plus Chemotherapy — camrelizumab+chemotherapy
  Arms: Arm A
Drug: placebo+chemotherapy — placebo+chemotherapy
  Arms: Arm B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of camrelizumab (an engineered anti-programmed death-ligand 1 [PD-1] antibody) plus chemotherapy vs placebo plus chemotherapy as neoadjuvant therapy in participants with triple negative breast cancer (TNBC). Participants will be randomized in a 1:1 ratio to Arm A (camrelizumab +chemotherapy) or Arm B (placebo + chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* ECOG Performance Status of 0-1.
* Early or locally advanced, histologically documented TNBC (absence of HER2, ER, and PR expression).
* Tumor stage: II-III.
* Adequate hematologic and organ function.
* Must be willing to use an adequate method of contraception for the course of the study.

Exclusion Criteria:

* Has a history of breast cancer.
* Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
* Has received prior chemotherapy, targeted therapy, and radiation therapy within the past 12 months.
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death - ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4].
* Has a diagnosis of immunodeficiency or autoimmune diseases.
* Has received any form of immunosuppressive therapy within 4 weeks prior to the first dose of study treatment.
* Severe pulmonary or cardiac disease.
* Known active hepatitis C virus, or known active hepatitis B virus.
* History of organ or bone marrow transplantation.
* Pregnant or breast-feeding women.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery. | Up to approximately 24 weeks

SECONDARY OUTCOMES:
Event-free Survival (EFS) as assessed by Investigator. | At least 2 years
  EFS is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Disease-free Survival (DFS) as assessed by Investigator | At least 2 years
  DFS is defined as the time from surgery to any of the following events: local or distant recurrence, or death due to any cause.
Distant Disease-free Survival (DDFS) as assessed by Investigator | At least 2 years
  DDFS is defined as the time from surgery to distant recurrence, or death due to any cause.
Objective response rate (ORR) in accordance with RECIST v1.1 | Up to approximately 24 weeks
  Number of responders Assessed by Modified Response Evaluation Criteria In Solid Tumours (RECIST v1.1) for target lesions assessed by MRI.
Percentage of Participants with Adverse Events (AEs) | Up to approximately 67 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen L, Li H, Zhang H, Yang H, Qian J, Li Z, Ren Y, Wang S, Fu P, Yang H, Liu Y, Sun J, Nie J, Lei R, Yao Y, Zhang A, Wang S, Ma X, Ouyang Z, Yang H, Wu SY, Cao SW, Wang K, Jiang A, Ouyang Q, Pang D, Wei L, Zha X, Shen Y, Qu X, Wu F, Zhu X, Wang Z, Fan L, Shao ZM. Camrelizumab vs Placebo in Combination With Chemotherapy as Neoadjuvant Treatment in Patients With Early or Locally Advanced Triple-Negative Breast Cancer: The CamRelief Randomized Clinical Trial. JAMA. 2025 Feb 25;333(8):673-681. doi: 10.1001/jama.2024.23560. PMID 39671272